CLINICAL TRIAL: NCT05549544
Title: Clinical Efficacy of Left Bundle Branch Area Pacing for Patients With Permanent Atrial Fibrillation and Heart Failure ：A Multi-center Randomized Controlled Trial
Brief Title: Clinical Efficacy of Left Bundle Branch Area Pacing for Patients With Permanent Atrial Fibrillation and Heart Failure
Acronym: LBBAP-AFHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xiaohan Fan, Professor, MD, PhD, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-1704
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Left Bundle Branch Area Pacing; Biventricular Pacing; Heart Failure; Permanent Atrial Fibrillation
Keywords: Left Bundle Branch Area Pacing; Permanent Atrial Fibrillation; Heart Failure; Biventricular Pacing
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBBAP group (Experimental): Device: Left bundle branch area pacing(LBBAP) LBBAP is a novel physiological pacing form for ventricular pacing. In patients who received LBBAP, the pacing lead will be placed at the left bundle branch area to achieve a narrow-paced QRS duration.
  Interventions: Device: Left bundle branch area pacing
- BiVP group (Active Comparator): Device: Biventricular pacing (BiVP) Biventricular pacing is the traditional pacing modality for patients with heart failure. For BiVP, one pacing lead was placed in the coronary sinus, named LV lead, and another lead was placed in the right ventricule.
  Interventions: Device: Biventricular pacing

INTERVENTIONS:
Device: Left bundle branch area pacing — Left bundle branch area pacing is a novel physiological pacing modality and is reported to be feasible and safe in patients with heart failure and left bundle branch block.
  Arms: LBBAP group
Device: Biventricular pacing — Biventricular pacing is a widely-established modality to treat heart failure in patients with heart failure
  Arms: BiVP group

SUMMARY:
This is a multicenter, randomized controlled study. This study aims to compare the clinical efficacy of LBBAP with traditional biventricular pacing in patients with permanent atrial fibrillation and heart Failure

DETAILED DESCRIPTION:
LBBAP-AFHF is a prospective, multicenter, randomized controlled trial that is designed to determine whether left bundle branch area pacing (LBBAP) may show superiority of improved LV function as compared with traditional biventricular pacing (BiVP) in patients with permanent atrial fibrillation and heart failure (LVEF<50%) who receive atrioventricular nodal ablation due to fast ventricular rate or require high percentage of ventricular pacing due to slow ventricular rate. The primary endpoint of this trial is the change in the LVEF at 6 months after device implantation from baseline. A CRT-P/D device would be implanted and LBBAP lead would be connected to the RA port and LV lead to the LV port. Patients who receive successful LBBAP and BiVP simultaneously during the procedure would be 1:1 randomized to LBBAP or BiVP group after the procedure by device programming. Patients will be followed at 3 and 6 months post-discharge for LVEF and other echographic parameters (including LVESV, response rate), and rehospitalization for heart failure or all-cause death.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged more than 18 years old
* Patients diagnosed with heart failure (LVEF<50%) and have received optimal medical therapy for at least 3 months
* Patients with permanent atrial fibrillation (QRS duration <130ms) which need ventricular pacing, including:

  1. LVEF<50%, NYHA II-IV, drug-refractory atrial fibrillation with the fast ventricular rate, planned atrioventricular nodal ablation due to 1). anticipated low success rate of atrial fibrillation catheter ablation or 2). patients refused to receive catheter ablation or 3). refused to receive another catheter ablation after a previous history of failed procedures
  2. LVEF<50%, NYHA II-IV, atrial fibrillation with slow ventricular rate, anticipated ventricular pacing burden ≥ 40%
* Written informed consent was provided

Exclusion Criteria:

* expected survival time is less than 12 months
* Prior history of mechanical tricuspid valve replacement and/or congenital heart disease (including dextrocardia, transposition of the great arteries, single left persistent left superior vena cava, etc.)
* Plan for PCI or CABG due to unstable angina or myocardial infarction in 3 months
* Surgery is required within 1 year due to severe structural heart disease
* Pregnancy, planned pregnancy or heart transplant
* Prior history of HCM and/or ventricular septal defect repair, who are unlikely to achieve successful LBBAP procedure.
* Failure of lead placement due to abnormal anatomy of the coronary sinus or enlarged right atrium, which makes it unable to switch from one pacing modality to another

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ΔLVEF between baseline and six months post-discharge | Six months after device implantation
  ΔLVEF：change in LVEF between baseline and six months after procedure

SECONDARY OUTCOMES:
The immediate success rate of the LBBAP procedure | 1 weeks
  Successful LBBAP procedure is identified according to ECG and intracardiac ECG electrogram (IEGM) during the procedure. All LBBAP procedures will be categorized as selective left bundle branch pacing (S-LBBP), non-selective left bundle branch pacing(NS-LBBP), or left ventricular septal pacing (LVSP).
The rate of procedure and Device related complications | 6 months
  Procedure complications include pneumothorax, hemothorax, and air embolism. Device related complications include lead and pocket complications
ΔLVEDD between baseline and six months post-discharge | 6 months
  ΔLVEDD：change in LVEDD between baseline and six months after procedure between two groups
ΔLVEDV between baseline and six months post-discharge | 6 months
  ΔLVEDV：change in LVEDV between baseline and six months after procedure between two groups
The echocardiographic response rate of LVEF increase ≥5% | 6 months
  the percentage of patients with change of LVEF ≥5% at 6 month from baseline
The changes of NT-proBNP betwen baseline and 6 months post-discharge | 6 months
  The changes of NT-proBNP betwen baseline and 6 months post-discharge
Composite incidence rate of all-cause mortality and/or hospitalization for heart failure | 6 months
  All-cause death: including cardiovascular and non-cardiovascular deaths. Hospitalization for heart failure: an unplanned outpatient or emergency department visit or inpatient hospitalization in which the patient presented with signs and symptoms consistent with heart failure and required medication therapy.
The echocardiographic response rate of LVEF increase ≥15% | 6 months
  an increase in LVESV ≥15% during follow-up at 6 month compared with baseline
The rate of ΔLVESV ≥15% between baseline and six months post-discharge | 6 months
  the percentage of patients with change of ΔLVESV ≥15% at 6 month from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohan Fan, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (5):
- China (5):
  - Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The first affiliated hospital of Nanjing medical university, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No